CLINICAL TRIAL: NCT07160270
Title: Neuropathy in Waldenström's Macroglobulinemia: Pathophysiology, Prognosis and Treatment
Brief Title: This Study Aims to Clarify the Prevalence and Characteristics of Neuropathy, Along With Associated Paraclinical Findings in Patients With Waldenström's Macroglobulinemia (WM) in a Cohort of WM Patients to Optimize the Diagnostic Process
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Morten Müller Aagaard, Medical doctor, Rigshospitalet, Denmark
Other Study IDs: H-23064477
Record Dates: First submitted 2025-06-02; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Waldenstrom Macroglobulinaemia; Peripheral Neuropathies
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — For patients included in the study with verified peripheral neuropathy and no other known cause than the association to Waldenströms Macroglobulinemia will be offered a genetic test for hereditary neuropathies though whole genome sequencing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuropathy associated to Waldenström's Macroglobulinemia

SUMMARY:
Neuropathy severely reduces patients' quality of life due to sensory loss, chronic neuropathic pain, and loss of mobility of arms and legs. Given the diverse origins of neuropathy, it is critical to identify its specific causes, particularly when effective treatments are available. Neuropathy is a frequent morbidity in Waldenström's macroglobulinemia (WM), a specific type of lymphoma caused by infiltration of clonal lymphoplasmocytic B cells in the bone marrow with the presence of IgM paraprotein. WM associated neuropathy is largely undescribed. The few existing studies are mostly retrospective indicating the neuropathy has a heterogenic pathophysiology and diverse clinical appearance from mild sensory neuropathy to aggressive with loss of ambulation and development of chronic neuropathic pain within weeks to months.

With treatment of WM the speed of the disease progression including the related neuropathy can be halted. Few studies and clinical experience indicate that the nerve damage induced by WM might remit if treatment is initiated early in the course of the disease. Thus, there is need for timely interventions to reduce chronic disabilities. However, even for an experienced neurologist, it can be difficult to identify whether the neuropathy is caused by WM or other causes where treatment is not indicated.

This project aims to investigate the prevalence and underlying mechanisms of neuropathy in patients with WM to help speed up the diagnostic process and thus help slow down the irreversible nerve damage that these patients experience.

DETAILED DESCRIPTION:
Methods

Study design: Cross-sectional observations study

Outcome:

Prevalence: Determining how many WM patients have neuropathy.

Characterization: Identification of clinical subtypes of WM associated neuropathy and their symptoms.

Biomarkers: Establishing relevant biomarkers (e.g., neurofilament light chain) to diagnose and predict neuropathy outcome.

We have already identified all patients with an active diagnosis of Waldenström Macroglobulinemia followed at the Department of Haematology at Rigshospitalet in august 2024. All patients have been screened with a questionnaire designed to identify signs of neuropathy. If probable symptoms of neuropathy the patients will be examined in the Department of Neurology. Almost 600 patients has been invided. 100 patients have symptoms fulfilling the criteria for probable neuropathy. With expect 90 patients patients in total to undergo clinical examination. Neuropathy will be clinically classified and confirmed with a nerve conduction study (ENG). Patient with neuropathy associated to WM will be further investigated with blood samples and lumbar puncture. The study duration will be one year, where we expect all participants to have gone through questionnaire, clinical examination, nerve conduction study and paraclinical tests. The follow up period will be for 3 years.

Clinical examination will be done by the responsible investigator Morten Müller Aagaard, MD.

Methodes include:

1. Clinical examination

   Neurological examination by a trained physician within the field of neuropathy.
2. Nerve conduction study (ENG)

   Paraclinical test of the sensory- and motornerves of the peripheral nervous system.
3. Questionnaires: I-RODS, FES-I, COMPASS 31, FSS and 5Q-5D
4. Blood samples

   The blood samples will be analysed with a standard polyneuropathy panel (liver, blood sugar/diabetes, kidney and hematologic markers e.g. interleukin-6, immunoglobulin A, G and M, kappa/lambda-chains and M-protein).

   Additionally the samples will be analysed for paraneoplastic antibodies, marker of neurodegenerative processes (e.g. neurofilament), rheumatologic markers (SSA, SSB, cryoglobulin, SR), and infection disorders as hepatitis b + c antibodies and HIV. In collaboration with department of immunology we also want to examine samples for complement activity and inflammation markers including cytokines.

   Whole genome squencing (WGS) for inherited neuropathies.
5. Cerebrospinal fluid

Cerebrospinal fluid will be examined with standard tests (erythrocytes, leucocytes, glucose, protein, neurofilament light polypeptide, borrelia, flowcytometry, cytology, and CXCL13)

The study duration will be 1 year with extra follow up for 3 years.

Statistics

The study is designed as a cross-sectional observation study describing WM associated neuropathy. The prevalence of neuropathy associated to WM will be estimated. Non-responders will be classified as missing data at random. In addition, sensitivity analyses will be conducted where the prevalence of neuropathy in non-responders will be varied within reasonable range and combined with information from the responders. Data will be processed using standard descriptive statistics, comparing results with normative reference values. Differences between WM patients and normal material will be analysed using t-tests, with p-values <0.05 considered statistically significant. The types of neuropathies, defined through electrophysiological and clinical phenotypes will undergo subgroup analyses based on group sizes. Statistical differences in clinical outcomes and biomarkers will be examined using ANOVA tests.

Impact

1. Clinical Understanding

   Enhanced Knowledge: The study will improve understanding of the prevalence, types, and pathophysiology of neuropathy associated with WM, leading to better recognition of the condition among healthcare providers.

   Treatment Guidelines: Establish clinical markers that may contribute to initiating or intensifying treatment for neuropathy associated with WM.
2. Patient Management

   Improved Diagnosis: Identification of specific biomarkers and clinical indicators will facilitate earlier and more accurate diagnoses of neuropathy, allowing for timely intervention.

   Optimal Monitoring: Contributing to better surveillance and management of WM regarding development of neuropathy in clinical practice.

   Tailored Treatments: Insights into which patients are likely to benefit from specific treatments can lead to studies about more personalized and effective treatment strategies.
3. Quality of Life

Functional Preservation: Addressing neuropathy early will lead to more rapid interventions both treatment and focus on the disabilities. Thus, patients may experience better maintenance of their mobility and daily functioning, thereby improving their overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Waldenström's Macroglobulinemia with symptoms of peripheral neuropathy for further clinical investigation.

Exclusion Criteria:

* Investigated with no sign of peripheral neuropathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Active diagnose of Waldenström's Macroglobulinemia under follow-up or has been followed at Rigshospitalet Department of Hematology.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of peripheral neuropathy associated to Waldenström Macroglobulinema (WM) | From enrollment from August 2024 and new diagnosed patients with WM and symptoms of neuropathy refered to the neuromuscular clinic until July 2025.
  The prevalence will be calculated by screening WM patients with a questionnaire designed specific for the research project to identify possible peripheral neuropathy. Patients with possible peripheral neuropathy will be clinical examined to either positiv og negative for peripheral neuropathy and confirmed by nerve conduction study. The prevalence will be the amount of patient with polyneuropathy in the population of investigated patientes with WM.

SECONDARY OUTCOMES:
Disability of WM associated polyneuropathy | Investigation during one year with follow up for 3 years
  The severity of WM associated neuropathy will be assesed by neuropathy scores - INCAT disability score (a scale of 0-10 with higher scores indicating greater disability.)
  * MRC 80 sum score (0-80. Lower score indicating more severe paralysis)
  * INCAT sensory sum score (0-20 with with higher scores indicating greater sensory abnormalities)
  * Modified Rankin scale: numbered 0 to 6, with higher scores indicating greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet Blegdamsvej., København Ø, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buske C, Castillo JJ, Abeykoon JP, Advani R, Arulogun SO, Branagan AR, Cao X, D'Sa S, Hou J, Kapoor P, Kastritis E, Kersten MJ, LeBlond V, Leiba M, Matous JV, Paludo J, Qiu L, Tam CS, Tedeschi A, Thomas SK, Tohidi-Esfahani I, Varettoni M, Vos JM, Garcia-Sanz R, San-Miguel J, Dimopoulos MA, Treon SP, Trotman J. Report of consensus panel 1 from the 11th International Workshop on Waldenstrom's Macroglobulinemia on management of symptomatic, treatment-naive patients. Semin Hematol. 2023 Mar;60(2):73-79. doi: 10.1053/j.seminhematol.2023.03.005. Epub 2023 Mar 29. PMID 37099027
- [Background] D'Sa S, Kersten MJ, Castillo JJ, Dimopoulos M, Kastritis E, Laane E, Leblond V, Merlini G, Treon SP, Vos JM, Lunn MP. Investigation and management of IgM and Waldenstrom-associated peripheral neuropathies: recommendations from the IWWM-8 consensus panel. Br J Haematol. 2017 Mar;176(5):728-742. doi: 10.1111/bjh.14492. Epub 2017 Feb 15. PMID 28198999
- [Background] Treon SP, Hanzis CA, Ioakimidis LI, Patterson CJ, Hunter ZR, Brodsky PS, m.fl. Clinical characteristics and treatment outcome of disease-related peripheral neuropathy in Waldenstrom's macroglobulinemia (WM). J Clin Oncol. 20. maj 2010;28(15_suppl):8114-8114.
- [Background] Hanewinckel R, Drenthen J, van Oijen M, Hofman A, van Doorn PA, Ikram MA. Prevalence of polyneuropathy in the general middle-aged and elderly population. Neurology. 2016 Nov 1;87(18):1892-1898. doi: 10.1212/WNL.0000000000003293. Epub 2016 Sep 28. PMID 27683845
- [Background] Dimopoulos MA, Kastritis E, Owen RG, Kyle RA, Landgren O, Morra E, Leleu X, Garcia-Sanz R, Munshi N, Anderson KC, Terpos E, Ghobrial IM, Morel P, Maloney D, Rummel M, Leblond V, Advani RH, Gertz MA, Kyriakou C, Thomas SK, Barlogie B, Gregory SA, Kimby E, Merlini G, Treon SP. Treatment recommendations for patients with Waldenstrom macroglobulinemia (WM) and related disorders: IWWM-7 consensus. Blood. 2014 Aug 28;124(9):1404-11. doi: 10.1182/blood-2014-03-565135. Epub 2014 Jul 15. PMID 25027391
- [Background] Castillo JJ, D'Sa S, Lunn MP, Minnema MC, Tedeschi A, Lansigan F, Palomba ML, Varettoni M, Garcia-Sanz R, Nayak L, Lee EQ, Rinne ML, Norden AD, Ghobrial IM, Treon SP. Central nervous system involvement by Waldenstrom macroglobulinaemia (Bing-Neel syndrome): a multi-institutional retrospective study. Br J Haematol. 2016 Mar;172(5):709-15. doi: 10.1111/bjh.13883. Epub 2015 Dec 21. PMID 26686858
- [Background] Viala K, Stojkovic T, Doncker AV, Maisonobe T, Lenglet T, Bruneteau G, Musset L, Neil J, Leger JM, Leblond V. Heterogeneous spectrum of neuropathies in Waldenstrom's macroglobulinemia: a diagnostic strategy to optimize their management. J Peripher Nerv Syst. 2012 Mar;17(1):90-101. doi: 10.1111/j.1529-8027.2012.00376.x. PMID 22462670
- [Background] Levine T, Pestronk A, Florence J, Al-Lozi MT, Lopate G, Miller T, Ramneantu I, Waheed W, Stambuk M, Stone MJ, Choksi R. Peripheral neuropathies in Waldenstrom's macroglobulinaemia. J Neurol Neurosurg Psychiatry. 2006 Feb;77(2):224-8. doi: 10.1136/jnnp.2005.071175. PMID 16421127
- [Background] Tomkins O, Leblond V, Lunn MP, Viala K, Weil DR, D'Sa S. Investigation and Management of Immunoglobulin M- and Waldenstrom-Associated Peripheral Neuropathies. Hematol Oncol Clin North Am. 2023 Aug;37(4):761-776. doi: 10.1016/j.hoc.2023.04.007. PMID 37385714
- [Background] Bibas M, Sarosiek S, Castillo JJ. Waldenstrom Macroglobulinemia - A State-of-the-Art Review: Part 1: Epidemiology, Pathogenesis, Clinicopathologic Characteristics, Differential Diagnosis, Risk Stratification, and Clinical Problems. Mediterr J Hematol Infect Dis. 2024 Jul 1;16(1):e2024061. doi: 10.4084/MJHID.2024.061. eCollection 2024. PMID 38984103
- [Background] Racine M. Chronic pain and suicide risk: A comprehensive review. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Dec 20;87(Pt B):269-280. doi: 10.1016/j.pnpbp.2017.08.020. Epub 2017 Aug 26. PMID 28847525
- [Background] Damci A, Schruers KRJ, Leue C, Faber CG, Hoeijmakers JGJ. Anxiety and depression in small fiber neuropathy. J Peripher Nerv Syst. 2022 Dec;27(4):291-301. doi: 10.1111/jns.12514. Epub 2022 Oct 7. PMID 36168866
- [Background] Streckmann F, Balke M, Cavaletti G, Toscanelli A, Bloch W, Decard BF, Lehmann HC, Faude O. Exercise and Neuropathy: Systematic Review with Meta-Analysis. Sports Med. 2022 May;52(5):1043-1065. doi: 10.1007/s40279-021-01596-6. Epub 2021 Dec 29. PMID 34964950
- [Background] Girach A, Julian TH, Varrassi G, Paladini A, Vadalouka A, Zis P. Quality of Life in Painful Peripheral Neuropathies: A Systematic Review. Pain Res Manag. 2019 May 23;2019:2091960. doi: 10.1155/2019/2091960. eCollection 2019. PMID 31249636